#### INFORMATION AND CONSENT FORM

For Adults and Parents/Guardians of Minor Participants

**Study Title:** A PHASE 3 RANDOMIZED, DOUBLE-BLIND, VEHICLE-CONTROLLED, PARALLEL GROUP STUDY OF A-101 TOPICAL SOLUTION APPLIED TWICE A WEEK IN SUBJECTS WITH COMMON WARTS

**Study #:** A-101-WART-301

**Sponsor:** Aclaris Therapeutics, Inc. **Study Doctor:** <<investigator>>

<<firm name>>

<<street address>>, <<city>>, <<state>><<zip>>

**Telephone Number:** <<000-000-0000>> **After Office Hours:** <<000-000-0000>>

The study doctor wants to know if you would like to be part of a research study.

If you have any questions about or do not understand something in this form, you should ask the study doctor or study staff. You should also discuss your participation with anyone you choose in order to better understand this study and your options.

Participating in a research study is not the same as getting regular medical care. The purpose of regular medical care is to improve your health. The purpose of a research study is to gather information.

When reading this form, please note that the words "you" and "your" refer to the person or child (persons under 18 years of age) participating in the study rather than to a parent/guardian who might sign this form on behalf of the person in the study.

#### WHAT IS THIS STUDY ABOUT?

You are being invited to participate in this research study because you have warts on your skin. The purpose of this research study is to test the safety and effectiveness of a new investigational drug, A-101 45% Topical Solution, that is applied only to the skin. An "investigational drug" is a drug that is being tested and is not approved for use in the United States by the U.S. Food and Drug Administration (FDA).

In addition, this study will compare A-101 45% Topical Solution with a placebo to see if using A-101 45% Topical Solution is better than using a placebo. The placebo is a solution that looks like A-101 45% Topical Solution but has no drug in it.

It is planned that about 500 people with common skin warts will be in this study.

Be aware that this form refers to A-101 45% Topical Solution as "study drug."

| Initials | Date |
|------------|-------------------|
| Version 1, | dated 27-JUL-2018 |
| Page 1 of | 13 |

### **HOW DOES A-101 45% TOPICAL SOLUTION WORK?**

A-101 45% Topical Solution contains hydrogen peroxide (H2O2). Hydrogen peroxide is a simple chemical combination of hydrogen and oxygen. H2O2 is commonly used in household products including chlorine-free bleaches, general-purpose cleaning agents and disinfectants, hair dyes and tooth-whitening products. In industry it is used in waste-water treatment and, at higher concentrations (greater than 30%), in bleaching paper pulp, and textiles. In medicine H2O2 is used at low concentrations (3%-6%) to cleanse wounds and as a topical antiseptic/disinfectant.

A-101 45% Topical Solution is being developed to remove common skin warts. This investigational drug containing H2O2 may remove warts due to its ability to dissolve the wart.

#### IS THERE ANYTHING ELSE I CAN DO FOR MY WARTS?

You do not have to be in this study to get help for your warts. Some other things you may be able to do are:

- Topical therapies such as acids (salicylic or trichloroacetic acids), available either overthe-counter or from a physician; cytotoxic therapies (topical podophyllin, cantharidin, 5fluorouracil, or bleomycin); topical immunomodulatory or immunotherapy (topical imiquimod, intralesional candida antigen, topical squaric acid dibutyl ester)
- Destruction of the warts by freezing (cryotherapy), electric current (electrosurgery), or scraping or cutting them off

You should discuss your alternatives to participating in this research with the study doctor or study staff. In addition, you may discuss your options with your regular health care provider.

## WHO IS PAYING FOR THIS STUDY?

A company called Aclaris Therapeutics, Inc., the sponsor of the study, is paying for this study.

<Quorum may add site-specific conflict-of-interest language to the form based on information the site reports to Quorum.>>

# WILL IT COST ANYTHING TO BE IN THIS STUDY?

There will be no charge to you for your participation in this study. The study drug, study-related procedures, and study visits will be provided at no charge to you or your insurance company.

# **HOW LONG WILL I BE IN THE STUDY?**

If you decide to be in this study and the study doctor says you can be in the study, your participation will last about 5 months and includes 13 visits to the study center.

If you decide to be in this study, you will first enter the study's screening period, which may last up to 13 days. If you continue your participation after the screening period, you will begin the study drug application period.

| Initials | Date |
|--------------|-------------------|
| Version 1, o | dated 27-JUL-2018 |

#### WHAT WILL HAPPEN DURING THIS STUDY?

If you decide to be in this study, you will have to stop any other wart therapies. This is known as a washout period. Your study doctor will tell you the length of any washout period needed. You will stop taking any of these therapies for the duration of your participation in the study.

You will be assigned by chance (like flipping a coin) to 1 of the following study groups:

- A-101 Topical Solution
- Placebo Solution (a solution that looks like A-101 45% Topical Solution but has no drug in it)

You have an equal chance of being in either of the study groups. Neither you nor the study doctor or study staff will be able to pick which study group you are in. You will not know and the study doctor or study staff will not know which study group you are in. The study doctor or study staff can find out if it is necessary to know for your health.

The study drug will be applied to up to 6 warts, which meet the requirement, twice a week for up to 8 weeks during visits 2 through 9. Participants between the ages of 12 and 17 years old will have their study drug applied once in the office by a parent of legal guardian in front of the study staff. The second application will be done at home by a parent or legal guardian as determined by the study doctor. Adult participants will be instructed by study staff how to self-apply study drug for the in-office treatment. The second application will be done at home by the participant as determined by the study doctor.

Study drug will be applied to each of the selected warts for about 15 seconds. Application with study drug at each visit may be repeated 3 times to each selected wart.

You will be given a study diary to record your applications of study drug at home.

While you are in the study, you must:

- Follow the instructions you are given.
- Come to the study center for all visits with the study doctor or study staff.
- Tell the study doctor or study staff about any changes in your health or the way you feel.
- Tell the study doctor or study staff if you want to stop being in the study at any time.
- Avoid scrubbing or irritating the warts being dosed you may continue your regular skin care products.
- Avoid excessive sun exposure to the warts being dosed.

## What happens when I come for study visits?

After you sign this form, the study doctor or study staff will do the things listed below when you come in for study visits.

# Visit 1 (Screening)

- **Demographic Questions:** You will be asked to give personal information, such as your name, date of birth, race, etc.
- **Health and Medication Questions:** You will be asked about your health, your medical history, and the medications you take.
- **Vital Signs:** Your blood pressure, heart rate, breathing rate, temperature, height and weight will be measured.
- Wart Assessment: Your skin will be assessed for warts. The study doctor will identify up to 6 common warts to be dosed with study drug. The warts will be measured.
- **Blood Testing:** Blood samples will be taken for routine laboratory evaluation.
- **Skin Type:** Your skin type will be assessed based on its shade/color.
- Photography: Photographs of your dosing areas (of the selected warts and nearby skin) will be taken throughout the study to document the location and status of the warts. These photographs may be used for research purposes related to the study and for presentation at the FDA, at scientific meetings, for scientific publications, for general corporate purposes, and may be used for marketing purposes. Your identity will not be revealed in these photographs. For example, if you have a distinctive birthmark or tattoo that is included in the photograph, the sponsor will take measures to digitally blur that feature from the photographs. If you decline to have these pictures taken, you will not be allowed to participate in this study.
- Subject Instruction Sheet: You will be given a written instruction sheet.

# Visit 2/ Day 1

- **Health and Medication Questions:** You will be asked about any changes to your health or medications.
- Wart Assessment: The common warts identified at Visit 1 will be looked at and measured by the study doctor.
- Review of Inclusion and Exclusion Criteria: The study doctor will confirm that you continue to meet all inclusion and no exclusion criteria.
- **Photography:** The warts will be photographed before study drug application.
- **Study Drug Application:** Study drug will be applied to the common warts identified by the study doctor.
- Evaluation of Application Area: The areas where study drug is applied will be examined for local skin reactions before study drug application. You will be asked about any stinging/burning or itching in those areas before study drug application.
- Subject Instruction Sheet: Your study instructions will be reviewed with you.

# <u>Visits 3 (Day 8), 4 (Day 15), Visit 5 (Day 22), Visit 6 (Day 29), Visit 7 (Day 36), and Visit 8 (Day 43)</u>

 Health and Medication Questions: You will be asked about any changes to your health or medications.

- Wart Assessment: The common warts will be looked at and measured by your study doctor.
- **Photography:** The common warts will be photographed at visit 4 and visit 6 only.
- **Study Drug Application:** Study drug will be applied to common warts during the inoffice visit as determined by the study doctor. The second weekly application of drug may be done home if the study doctor thinks you need another application.
- Evaluation of Application Area: The areas where study drug is applied will be examined for local skin reactions before study drug application. You will be asked about any stinging/burning or itching in those areas before study drug application, if applicable.
- Subject Instruction Sheet: Your study instructions will be reviewed with you.

# Visit 9/Day 50 (End of Dosing)

- Health and Medication Questions: You will be asked about any changes to your health or medications.
- Vital Signs: Your blood pressure, heart rate, breathing rate, and temperature will be measured.
- Wart Assessment: The common warts will be looked and measured by the study doctor.
- **Photography:** The common warts will be photographed.
- **Study Drug Application:** Study drug will be applied to common warts during the inoffice visit as determined by the study doctor. The second weekly application of study drug may be done at home if the study doctor thinks you need another application.
- Evaluation of Application Area: The areas where study drug is applied will be examined for local skin reactions before study drug application. You will be asked about any stinging/burning or itching in those areas before study drug application, if applicable.
- Subject Instruction Sheet: Your study instructions will be reviewed with you.

# Visits 10 (Day 60), 11 (Day 78), and 12 (Day 106) - Follow-up Visits

- **Health and Medication Questions:** You will be asked about any changes to your health or medications.
- Photography: The common warts will be photographed at Visit 10, Visit 11, & Visit 12.
- Wart Assessment: The common warts will be looked at and measured by the study doctor.
- Evaluation of Application Area: The areas where study drug was applied will be examined for local skin reactions. You will be asked about any stinging/burning or itching in those areas.
- Subject Instruction Sheet: Your study instructions will be reviewed with you.

# Visit 13 – End of Study

 Vital Signs: Your blood pressure, heart rate, breathing rate, and temperature will be measured.

- **Blood Testing:** Blood samples will be taken for routine laboratory evaluation.
- **Photography:** The common warts will be photographed.
- Wart Assessment: The common warts will be looked at and measured by the study doctor.
- Evaluation of Application Area: The areas where study drug was applied will be examined for local skin reactions. You will be asked about any stinging/burning or itching in those areas.

# **Early Discontinuation Visit**

If you decide you do not want to be in the study anymore for any reason, the procedures for Visit 13 will be completed.

#### WILL BEING IN THIS STUDY HELP ME?

The study drug may help your warts, but there is no guarantee that being in this study will help you. Your warts might not get better or may even get worse while you are in this study. You may get placebo, which has no drug in it. Information from this study might help researchers come up with medications to help others in the future.

## WHAT ARE THE RISKS TO ME IF I AM IN THIS STUDY?

Ask the study doctor if you have questions about the signs or symptoms of any side effects that you read about in this consent form. Hydrogen peroxide has been used in people for other reasons, and when it is applied topically the common adverse effects include:

- Temporary discomfort in the dosing area (burning, stinging and/or itching)
- · Temporary redness in the dosing area
- Temporary and reversible whitening (NOT BLEACHING) of the skin
- Blistering
- Bleaching of the hair within the dosing area.

In a previous study of subjects using hydrogen peroxide the side effects seen included:

- Stinging or burning sensation at the study drug application site
- Mild discomfort at the site

While not a side effect, H2O2 may bleach clothing that overlies the application area or comes in contact with the study drug.

Precaution: The study drug is a high-strength hydrogen peroxide product. High strength hydrogen peroxide products may cause serious harm or death if ingested. High strength hydrogen peroxide products are highly corrosive, and the FDA considers the substance to be dangerous. A-101 hydrogen peroxide should only be applied topically as indicated for skin warts.

It is possible that using A-101 may change how your regular medications, vaccines, or supplements work. It is very important that you tell the study doctor about any medications, supplements, or vaccines before you take them during the study.

Please tell the study doctor or study staff right away if you have any side effects. Please tell them if you have any other problems with your health or the way you feel during the study, whether or not you think these problems are related to the study drug.

If you feel that A-101 45% topical solution has come in contact with your eyes, mouth or nose, tell your study doctor immediately. Serious eye problems may happen if the solution gets into your eyes. Eye problems may include, pain, swelling, redness, irritation and in some cases, blindness.

# Could I have an allergic reaction?

All topical drugs have a potential risk of an allergic reaction, which could result in a rash (red or rough skin) or a worse skin reaction at the area of application.

# What if I am using placebo instead of A-101 during the study?

Some people in the study will get placebo instead of A-101 45% hydrogen peroxide. Placebo is a substance that looks like A-101 topical solution but has no hydrogen peroxide in it. If you use placebo during the study, it is possible that your warts may get worse. Please ask the study doctor or study staff if you have any questions about placebo.

## If I stop my regular medication, therapy, or supplements what are the risks?

If you stop your regular medication, therapy, or supplements to be in the study, your warts symptoms might come back or get worse. Please tell the study doctor or study staff right away if you have any problems when you stop or change your regular medication, therapy, or supplements.

## What are the risks of giving blood for this study?

The study doctor or study staff will take your blood by sticking a needle in your arm. Some problems you might have from this are:

- pain
- bruising
- dizziness
- infection

### Unknown risks

It is possible that you could have problems and side effects of A-101 topical solution that nobody knows about yet, which could include your warts getting worse.

# Loss of confidentiality

There is a risk of loss of confidentiality of your information. You will read more about the protection of your information later in this form. Please ask the study doctor or study staff if you would like to know more about how your information will be protected while you are in this study.

#### WILL I RECEIVE ANY NEW INFORMATION DURING THE STUDY?

If the study doctor or study staff learns any new information that might change your mind about continuing in the study, the study doctor or study staff will tell you about it.

## WHAT IF I GET HURT OR SICK WHILE I AM IN THIS STUDY?

If, during the course of this study, any injury occurs to you as a direct result of the administration of the study drug or properly performed procedures, the Sponsor agrees to pay all medical expenses necessary to treat such injury: 1) to the extent you are not otherwise reimbursed by medical insurance; 2) provided you have followed the directions of the study doctor.

Compensation for any injury which occurs to you as a direct result of the administration of the study drug or poorly performed procedures by the study doctor or study staff, will be paid after the Sponsor receives all appropriate documentation and completes its review, to its satisfaction, of all documentation regarding your claim for injury.

You will not lose any of your legal rights or release the Sponsor, the study doctor, the study staff, or study site from liability for negligence or intentional misconduct by signing this consent form.

There are no plans to provide financial compensation for such things as lost wages, disability or discomfort due to injury.

Be aware that your health care payer/insurer might not cover the costs of study-related injuries or illnesses.

#### WILL I RECEIVE PAYMENT?

<< Quorum will add site-specific compensation language to the form based on information the site reports to Quorum.>>

#### DO I HAVE TO BE IN THIS STUDY?

Your participation in this study is voluntary. You can decide not to be in the study and you can change your mind about being in the study at any time. There will be no penalty to you, and you

| Initials | Date |
|--------------|------------------|
| Version 1, d | ated 27-JUL-2018 |

won't lose any benefits you are entitled to. If you want to stop being in the study, tell the study doctor or study staff.

The study doctor or study staff or sponsor can remove you from the study at any time, even if you want to stay in the study. This could happen if:

- The study doctor or study staff believes it is best for you to stop being in the study.
- You do not follow directions about the study.
- The sponsor stops the study for any reason.

If you stop being in the study early, the study doctor or study staff may ask you some questions about being in the study. The study doctor or study staff may ask you to participate in some procedures or tests to help you leave the study safely and/or to collect more information for the study. If you leave the study, the study doctor and study staff will still be able to use your information that they have already collected.

## **HOW WILL MY INFORMATION BE KEPT CONFIDENTIAL?**

Your identity will be protected as required by law and according to any policies the study center or sponsor may have. Be aware that your study records (which include your medical records, your signed consent form, and other information) will be shared as needed for the study. For example, the U.S. Food and Drug Administration (FDA), Aclaris Therapeutics, Inc. and Quorum Review (a group of people who review research studies to protect the rights and welfare of research participants) may look at your study and medical records.

Your blood samples will not be labeled with your name or other directly identifying information. Your samples will have a code instead. The list that matches the code with your name will be stored separately from your samples. Your samples will be kept only until we are able to complete the tests described in this form, and then your samples will be destroyed. If you change your mind later, be aware that your samples may or may not be withdrawn from the research, depending on the sponsor's policies. You can ask the study doctor or study staff about this.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## WHO CAN I TALK TO ABOUT THIS STUDY?

In the event of an emergency, dial 911 immediately.

If you require emergency care, be sure to tell the emergency care provider about your participation in this study. Contact the study doctor or study staff as soon as possible.

You can ask questions about the study at any time. You can call the study doctor or study staff at any time if you have any concerns or complaints. You should call the study doctor or study staff at the phone number listed on page 1 of this form if you have questions about the study procedures, study payment, or if you get hurt or sick during the study.

| Initials | Date |
|-------------|-------------------|
| Version 1, | dated 27-JUL-2018 |

Quorum Review reviewed this study. Quorum Review is a group of people who review research studies to protect the rights and welfare of research participants. Review by Quorum Review does not mean that the study is without risks. If you have questions about your rights as a research participant, if you are not able to resolve your concerns with the study doctor or study staff, if you have a complaint, or if you have general questions about what it means to be in a research study, you can call Quorum Review or visit the Quorum Review website at www.QuorumReview.com.

Quorum Review is located in Seattle, Washington.

Office hours are 8:00 AM to 5:00 PM Pacific Time, Monday through Friday. Ask to speak

with a Research Participant Liaison at 888-776-9115 (toll free).

## HOW WILL MY INFORMATION BE USED AND SHARED FOR THIS STUDY?

This section explains who will use and share your health information if you agree to be in this study. You must authorize this use and sharing of your information by signing this form or you cannot be in the study.

The study doctor and study staff will collect, use, and share health information about you, including any information needed to do the study and other identifying information about you, such as your name, address, phone number, or social security number. The information used and shared will include:

- information from your medical records
- information collected about you during the research including study visits, progress notes, tests, procedures, photographs, etc.

Your information may be used and shared with these people for the following purposes:

- The study doctor and study staff to conduct this research.
- The sponsor, Aclaris Therapeutics, Inc.; people who work with or for the sponsor; and other researchers involved in this study. These people will use your information to review the study, to check the safety and results of the study, and to seek government approval of A-101 45% Topical Solution.
- Others required by law to review the quality and safety of research, including the FDA, Department of Health and Human Services, Office for Human Research Protections, other government agencies in the United States and other countries, and Quorum Review.

After your information is shared with the people and companies listed above, the law may not require them to protect the privacy of your information. To maintain the integrity of this research, you might not have access to any health information developed as part of this study until it is completed. At that point, you generally would have access to your health information.

You can cancel your authorization to use and share your information at any time by writing a letter to the study doctor. If you cancel your authorization, you will not be able to continue in the study. If you cancel your authorization, the study doctor and study staff will still be able to use and share your information that they have already collected.

This authorization to use and share your information expires in 50 years.

| Initials | Date |
|--------------|-------------------|
| Version 1, o | dated 27-JUL-2018 |
| Page 10 of | 13 |

# REGULAR DOCTOR OR SPECIALIST NOTIFICATION OPTION

For your safety, you or the study doctor should tell your regular health care provider that you are in this study. This is recommended so that your primary care doctor may contact the study doctor if they have any concerns or questions about your care.

| 400101 | in they have any concerns or queetiene abou | at your ouro. |
|---|---|---|
| | se indicate below whether you want us to not<br>our participation in this study. | ify your regular doctor or your specialist |
| | Yes, I want the study doctor to inform my in this study: | regular doctor/specialist of my participation |
| Name | of Doctor | Phone |
| Name | of Doctor No, I do not want the study doctor to inform my participation in this study. | |
| _ | No, I do not want the study doctor to infor | |

### CONSENT

I have read this form, and I have been able to ask questions about this study. The study doctor or study staff has talked with me about this study. They have answered all my questions. I voluntarily agree to be in this study. I agree to allow the collection, use, and sharing of my information as described above.

By signing this form, I do not give up any of my legal rights. I will get a signed copy of this consent form. Printed Name of Participant Signature of Participant (if an Adult) Date << Quorum staff: Include the following for Indiana sites: In **Indiana**, you must complete the following information: Participant's Street Address Participant's City, State, ZIP>> If participant does not have the legal capacity to consent to his/her participation: I am the parent/guardian of the participant named above and I consent to his/her participation in this research study. I also authorize the collection, use and sharing of the participant's information. Printed Name of Parent/Guardian Signature of Parent/Guardian Date

Initials \_\_\_\_\_ Date \_\_\_\_ Version 1, dated 27-JUL-2018 Page 12 of 13

| I attest that the individual providing consent had enough tim<br>an opportunity to ask questions, and voluntarily agreed to p | |
|---|---|
| Printed Name of Person Explaining Consent | |
| Signature of Person Explaining Consent | Date |
| I attest that I or my representative discussed this study with | the individual providing consent. |
| Signature of Principal Investigator or Sub-Investigator | |